CLINICAL TRIAL: NCT00553280
Title: An Open-Label Extension Safety And Efficacy Study Of Pregabalin (CI-1008) For Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: A Long-Term Study To Evaluate Safety And Efficacy Of Pregabalin For Pain Associated With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081164
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2011-04

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pregabalin (Experimental)
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — Dosage: 150-600 mg/day (75-300 mg bid), oral administration, Treatment duration: 52 weeks

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the long-term use of pregabalin at doses up to 600 mg/day in patients with painful diabetic peripheral neuropathy who have completed 13 weeks of dosing in Study A0081163

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the 13-week treatment of painful diabetic peripheral neuropathy in Study A0081163.
* Patients must be able to understand and cooperate with study procedures and have signed a written informed consent prior to entering the study

Exclusion Criteria:

* Patients who experienced serious adverse events in the preceding study (A0081163) that were determined by the investigator or the study sponsor to be causally related to the study medication.
* Patients exhibiting treatment non-compliance in the preceding study (A0081163)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- Japan (27):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Date-shi, Fukushima
  - Pfizer Investigational Site, Nihommatsu, Fukushima
  - Pfizer Investigational Site, Shirakawa-shi, Fukushima
  - Pfizer Investigational Site, Sukagawa, Fukushima
  - Pfizer Investigational Site, Kamakura, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Matsumoto, Nagano
  - Pfizer Investigational Site, Ueda, Nagano
  - Pfizer Investigational Site, Beppu, Oita Prefecture
  - Pfizer Investigational Site, Yamada, Okayama-ken
  - Pfizer Investigational Site, Naha, Okinawa
  - Pfizer Investigational Site, Tomishiro, Okinawa
  - Pfizer Investigational Site, Urazoe, Okinawa
  - Pfizer Investigational Site, Hirano-ku, Osaka
  - Pfizer Investigational Site, Suminoe-ku, Osaka
  - Pfizer Investigational Site, Sunto-gun, Shizuoka
  - Pfizer Investigational Site, Oyama-shi, Tochigi
  - Pfizer Investigational Site, Arakawa City, Tokyo
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Ohta-ku, Tokyo
  - Pfizer Investigational Site, Shibuya-ku, Tokyo
  - Pfizer Investigational Site, Fukuoka
  - Pfizer Investigational Site, Ōita
  - Pfizer Investigational Site, Tokushima

REFERENCES:
- [Derived] Satoh J, Yagihashi S, Baba M, Suzuki M, Arakawa A, Yoshiyama T. Efficacy and safety evaluation of pregabalin treatment over 52 weeks in patients with diabetic neuropathic pain extended after a double-blind placebo-controlled trial. J Diabetes Investig. 2011 Nov 30;2(6):457-63. doi: 10.1111/j.2040-1124.2011.00122.x. PMID 24843530
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081164&StudyName=A%20Long-Term%20Study%20To%20Evaluate%20Safety%20And%20Efficacy%20Of%20Pregabalin%20For%20Pain%20Associated%20With%20Diabetic%20Peripheral%20Neuropathy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-six (36) centers in Japan
Pre-assignment Details: Patients with pain associated with diabetic peripheral neuropathy who had completed the 13-week treatment phase in the preceding study (Study A0081163: NCT00553475), without any treatment-related serious adverse events or any compliance problems were eligible for the study.
Groups:
- Pregabalin: Participants initiated to take the study drug at a dose of 75 mg in the evening of Day 1, and then 150 mg/day (75 mg BID) for 1 week from Day 2. Thereafter, participants continued the treatment with pregabalin for 52 weeks, with the maximum doses of 300 mg/day (150 mg BID) for participants with low CLcr (30 < CLcr ≤ 60 mL/min) and 600 mg/day (300 mg BID) for participants with normal CLcr (CLcr > 60 mL/min). In consideration of safety and the effect on pain, the doses were adjusted by one step (150 mg/day) at each visit. Participants treated with pregabalin at the doses of 300 mg/day or higher ended the treatment after a 1-week dose reduction period.
Period: Overall Study
Arm/Group | Pregabalin
Started | 123
Completed | 97
Not Completed | 26
Not completed — Adverse Event | 19
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 123
Age, Customized [Number; unit: participants]
  < 18 years | 0
  18 - 44 years | 6
  45 - 64 years | 71
  >= 65 years | 46
Age, Customized [Mean (Standard Deviation); unit: years] | 61.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 100

OUTCOME MEASURES:

1. Primary Outcome: Summary of Adverse Events
Description: Number of participants with all causality adverse events, serious adverse events, severe adverse events, adverse events resulted in discontinuation, dose reduced or temporary discontinuation. Participants are counted only once per treatment in each row.
Time Frame: 53 weeks
Population: Safety analysis set: all participants who had received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 123
participants
  Participants with adverse events | 114
  Participants with serious adverse events | 21
  Participants with severe adverse events | 7
  Participants discontinued due to adverse events | 17
  Dose reduced or temporary discontinuation | 43

2. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Sensory Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Sensory score ranges from 0-33. Higher scores indicate more severe pain.
Time Frame: From baseline to 52 weeks or study discontinuation (Study Endpoint)
Population: Full analysis set. No imputations for missing data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 123
score on scale | -3.5 (5.1)

3. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Affective Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Affective score ranges from 0-12. Higher scores indicate more severe pain.
Time Frame: From baseline to 52 weeks or study discontinuation (Study Endpoint)
Population: Full analysis set. No imputations for missing data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 123
score on scale | -1.2 (2.4)

4. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Total Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Total score ranges from 0-45. Higher scores indicate more severe pain.
Time Frame: From baseline to 52 weeks or study discontinuation (Study Endpoint)
Population: Full analysis set. No imputations for missing data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 123
score on scale | -4.7 (6.8)

5. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Visual Analogue Scale Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Visual Analogue Scale Score ranges from 0-100 mm. Higher scores indicate more severe pain.
Time Frame: From baseline to 52 weeks or study discontinuation (Study Endpoint)
Population: Full analysis set. No imputations for missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin
Number analyzed (Participants) | 123
mm | -25.4 (26.4)

6. Secondary Outcome: Change From Baseline in Short-Form McGill Pain Questionnaire: Present Pain Intensity Scores
Description: The mean change from baseline in Short-Form McGill Pain Questionnaire Scores at study endpoint. Present pain intensity score ranges from 0-5. Higher scores indicate more severe pain.
Time Frame: From baseline to 52 weeks or study discontinuation (Study Endpoint)
Population: Full analysis set. No imputations for missing data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 123
score on scale | -0.7 (1.1)

ADVERSE EVENTS:
Time Frame: 53 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 21/123
Other Adverse Events (participants affected / at risk) | 101/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=123)
Atrioventricular block complete (Cardiac disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Cellulitis (Infections and infestations) | 2
Diabetic gangrene (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Blood glucose abnormal (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=123)
Diabetic retinopathy (Eye disorders) | 9
Visual acuity reduced (Eye disorders) | 7
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 8
Face oedema (General disorders) | 10
Oedema (General disorders) | 9
Oedema peripheral (General disorders) | 21
Nasopharyngitis (Infections and infestations) | 39
Contusion (Injury, poisoning and procedural complications) | 8
Fall (Injury, poisoning and procedural complications) | 14
Weight increased (Investigations) | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 29
Somnolence (Nervous system disorders) | 30
Eczema (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.